CLINICAL TRIAL: NCT01064596
Title: Fondaparinux Population Pharmacokinetic to Morbid Obese Patients in Post-operatory Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 0908104; 2009-016417-15 (EudraCT Number)
Record Dates: First submitted 2010-01-11; First posted 2010-02-08 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Morbid Obesity; Obesity; Surgery
Keywords: obesity; fondaparinux; surgery; anti-Xa activity
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4 blood samples to measure anti-Xa activity
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- blood sample: Patient with 4 blood samples to measure anti-Xa activity
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — patients with a fondaparinux treatment who have 4 blood samples during the 10 days following surgery

SUMMARY:
After bariatric surgery , thromboembolics complications are major cause of mortality. However, in obese patients, thromboprophylaxia is a controversy. Fondaparinux' efficacy is superior to HBPM, and is a good treatment for this population. Pharmacokinetics information with Fondaparinux in this population are rare.

DETAILED DESCRIPTION:
We proposed a bicentric study cohort of obese patients (BMI > 40 kg/m2) treated by 1 day injection of Fondaparinux 2.5 mg after bypass surgery. Anti-Xa activity of Fondaparinux will be measured 4 times during hospitalisation for each patient to realise a pharmacokinetic modelisation of Fondaparinux. Haemorrhage and thromboembolics events will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* requiring a bariatric surgery
* requiring an antithrombotics prophylaxis
* having a morbid obesity based on a BMI >40 kg/m2
* having signed the inform consent form

Exclusion Criteria:

* contra-indication to fondaparinux
* history of heparin induced thrombopenia (HIT)
* platelets < 100 G/l
* requiring an effective antithrombotic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obesity patients who need a bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To evaluate pharmacodynamics parameters of fondaparinux based on anti-Xa activity estimated by a non linear model at mixed effect of obese morbid patients following a bariatric surgery | 5 days

SECONDARY OUTCOMES:
To evaluate the incidence of symptomatic venous thromboembolics events (DVT and PE) between D5 and D10 and at 1month ± 10 days | D5
the incidence of major and clinically significative bleeding between D5 and D10 and at 1 month ± 10 days | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MISMETTI, MD, PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (3):
- France (3):
  - Assistance Publique - Hôpitaux de Paris, Paris
  - Clinique de la Mutualiste, Saint-Etienne
  - Chu de Saint-Etienne, Saint-Etienne